CLINICAL TRIAL: NCT00815919
Title: A Phase II Trial of Bortezomib (Velcade) Plus Prednisone for Initial Therapy of Chronic Graft Versus Host Disease
Brief Title: Bortezomib Plus Prednisone for Initial Therapy of Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-191
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: cGVHD; Velcade; bortezomib
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Bortezomib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Velcade (bortezomib) (Experimental)
  Interventions: Drug: bortezomib; Drug: Prednisone

INTERVENTIONS:
Drug: bortezomib — Given intravenously at a dose of 1.3 mg/m^2 once a week for the first four weeks of a five week cycle for a total of 3 cycles
  Other Names: Velcade
Drug: Prednisone — Taken orally once a day at a dose of 0.5-1 mg/kg. Dose reduction may be initiated after 1 cycle of therapy. A suggested taper is 10-25% every 1-2 weeks.

SUMMARY:
The purpose of this research study is to determine the effectiveness of bortezomib (Velcade) plus prednisone for treating chronic graft versus host disease (cGVHD) and the safety of this drug combination in this patient population. Chronic GVHD is a medical condition that may occur after allogeneic stem cell transplantation. The donor's immune system may recognize the participants body (the host) as foreign and attempt to "reject" it. Bortezomib has been used in other research studies, and information from those studies suggests that this drug may help to control the abnormal immune responses that underlie cGVHD.

DETAILED DESCRIPTION:
* Each treatment cycle lasts five weeks, during which time participants will come to the clinic to receive bortezomib intravenously once a week for the first 4 weeks. Prednisone will be taken orally on a daily basis and dose reduction may be initiated after 1 cycle of therapy.
* During all treatment cycles, participants will have the following: physical exam and blood work. At the end of cycle 3 (week 15) the participants cGVHD will be evaluated. These assessments may include an eye examination, a skin examination, a pulmonary function test and/or, a flexion assessment test.
* Participants will receive 3 cycles of bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic stem cell transplantation with myeloablative or non-myeloablative conditioning regimens
* 100 days or more past stem cell transplantation
* Recipients of matched or mismatched, related or unrelated adult donor stem cells
* Must have cGVHD requiring systemic therapy
* No addition or subtraction of other immunosuppressive medications. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug. However, if cGVHD occurs during a taper of immune suppression, the medication(s) may not be increased back up to therapeutic level, but will continue a the taper dose for the 15 week study duration
* Adequate bone marrow, hepatic and renal function as outlined in the protocol
* Does not require hemodialysis
* 18 years of age or older
* ECOG Performance Status of 0-2 or Karnofsky performance score of 70% or greater
* Life expectancy of more than 3 months

Exclusion Criteria:

* Systemic steroid therapy in the 4 weeks prior to enrollment
* Active malignant disease after transplantation. Complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy will not be considered in this category
* Active uncontrolled infection
* Peripheral neuropathy CTC Grade 1 (or greater) with pain in the 4 weeks before enrollment. Other neurological deficits must be reviewed with the study PI prior to study entry
* Myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Hypersensitivity to bortezomib, boron, or mannitol
* Female subject is pregnant or breast-feeding
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-12; Primary Completion 2012-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MBBS, DPhil, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade (Bortezomib): Prednisone : Taken orally once a day at a dose of 0.5-1 mg/kg. Dose reduction may be initiated after 1 cycle of therapy. A suggested taper is 10-25% every 1-2 weeks.
  Bortezomib : Given intravenously at a dose of 1.3 mg/m^2 once a week for the first four weeks of a five week cycle for a total of 3 cycles
Period: Overall Study
Arm/Group | Velcade (Bortezomib)
Started | 22
Completed | 18
Not Completed | 4
Not completed — Unrelated Fungal Infection | 1
Not completed — AML Relapse | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Velcade (Bortezomib)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 51 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate After a 15 Week Course of Bortezomib Plus Prednisone in Patients With cGVHD
Description: Participants had their cGVHD evaluated per NIH consensus criteria:
  Complete response: resolution of all reversible manifestations of cGVHD.
  Partial response: a decrease ≥ 1 point on a 3-point organ-specific scale or 2 points or more on a 10-point global scale without progression in any organ sites.
  Stable disease: no evidence of cGVHD response without evidence of progressive cGVHD.
  Progressive cGVHD: increase of ≥ 1 point on an organ-specific 3-point scale, addition of a new immunosuppressive agent prior to the completion of 15 weeks of combination therapy, or requirement an increase in the total daily dose of corticosteroids above a participant's baseline corticosteroid dose during the 15-week combined treatment period.
  Mixed response: a response in primary sites of cGVHD involvement but interval progressive cGVHD in other organs or sites.
  Responses were not scored for oral or ocular cGVHD, since topical therapies were permitted during the study.
Time Frame: Patients had their cGVHD assessed at Baseline and at 15 weeks or end of therapy
Measure: Number; unit: participants
Arm/Group | Velcade (Bortezomib)
Number analyzed (Participants) | 20
participants
  Participants with a complete response in cGVHD | 2
  Participants with an partial response in cGVHD | 14
  Participants with stable cGVHD | 1
  Participants with progressive cGVHD | 2
  Participants with mixed response | 1

2. Secondary Outcome: Proportion of Patients Tolerating >50% Steroid Dose Reduction After a 15 Week Course of Bortezomib Plus Prednisone in Patients With cGVHD
Description: The participants' total daily steroid dose was recorded at baseline and after a 15 week course of treatment. Starting at a dose of 0.5-1 mg/kg, dose reduction of steroids was permitted after 1 cycle of therapy. The suggested taper was 10-25% every 1-2 weeks. .
Time Frame: After 15 weeks of bortezomib plus prednisone therapy
Population: Of the overall 22 patients, 18 patients completed 3 cycles (15 weeks) of therapy
Measure: Number; unit: participants
Arm/Group | Velcade (Bortezomib)
Number analyzed (Participants) | 18
participants | 14

3. Secondary Outcome: The Toxicity of a 15 Week Course of Bortezomib Plus Prednisone in Patients With cGVHD
Description: Participants' toxicities were graded based on the CTCAE version 3.0. The toxicities were then given an attribution to the velcade treatment: unrelated, unlikely, possible, probable, definite.
Time Frame: Toxicities were collected from the start of treatment through 15 weeks of therapy or end of study treatmetn
Measure: Number; unit: participants
Arm/Group | Velcade (Bortezomib)
Number analyzed (Participants) | 22
participants
  Participants with >= Grade 3, unrelated/unlikely | 7
  Participants with >= Grade 3, possible | 1
  Participants with >= Grade 3, probable/definite | 0

4. Secondary Outcome: Proportion of cGVHD Patients Requiring Prednisone by 1 Year After Therapy
Description: Participants who were still being followed 1 year after the start of therapy had their prednisone dose recorded.
Time Frame: 1 year after the start of study treatment
Population: Participants who were still being followed 1 year after the start of therapy.
Measure: Number; unit: participants
Arm/Group | Velcade (Bortezomib)
Number analyzed (Participants) | 17
participants
  Participants still requiring prednisone | 11
  Participants off prednisone | 6

5. Secondary Outcome: Overall and cGVHD Progression-free Survival by 1 Year After Therapy
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Velcade (Bortezomib)
Number analyzed (Participants) | 22
percentage of participants
  2-year Cum-incidence of Non-relapse mortality | 14 [3 to 31]
  2-year Cum-incidence of malignant relapse | 14 [3 to 31]
  2 year progression-free survival | 73 [49 to 87]
  2-year Overall survival | 73 [49 to 87]

ADVERSE EVENTS:
Groups:
- Velcade (Bortezomib): Prednisone : Taken orally once a day. Dose reduction may be initiated after 1 cycle of therapy. A suggested taper is 10-25% every 1-2 weeks.
  bortezomib : Given intravenously once a week for the first four weeks of a five week cycle for a total of 3 cycles
Arm/Group | Velcade (Bortezomib)
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 7/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade (Bortezomib) (N=22)
Relapse AML (Blood and lymphatic system disorders) | 1 (1) — Patient died of relasped AML disease.
Infection (Infections and infestations) | 1 (1) — Patient died of an unrelated fungal infection
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade (Bortezomib) (N=22)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Neuropathy- sensory (Nervous system disorders) | 1 (1)
ALT-SGPT elevated (Metabolism and nutrition disorders) | 2 (2)
AST-SGOT elevated (Metabolism and nutrition disorders) | 2 (2)
Alkaline Phosphotase elevated (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes